CLINICAL TRIAL: NCT05088408
Title: Comparative Study Between Colonoscopy Bowel Preparation With Clear Liquids, With and Without Two Servings of High Energy Nutritional Supplement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clínica de Gastroenterologia (Other)
Collaborators: Nestlé Portugal SA (Unknown); Angelini Pharma Portugal, Unipessoal, Lda (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 01
Record Dates: First submitted 2021-07-10; First posted 2021-10-21 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Colonoscopy; Bowel Preparation

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Active Comparator): Bowel preparation as usual. Colonoscopy.
  Interventions: Other: Bowel preparation as usual.
- Dietary supplement (Experimental): Bowel preparation as usual plus two bottles of the dietary supplement Resource® Energy Apricot.
  Colonoscopy.
  Interventions: Dietary Supplement: Resource® Energy Apricot

INTERVENTIONS:
Dietary Supplement: Resource® Energy Apricot — Bowel preparation as usual plus two bottles of Resource® Energy Apricot (one day before the colonoscopy with no ingestion of solid foods, possibly with ingestion of clear liquids with or without sugar (such as tea or other transparent beverages without pulp, but not milk, yogurt, broth or gelatine), with ingestion of one bottle of 200 mL of the dietary supplement at 08:00 and the other at 12:00, and with ingestion of 275,84 g (4 sachets) of polyethylene glycol 3350 (Klean-Prep®) in 4 litres of water in 3 to 4 hours (250 mL every 15 minutes), starting at 18:00; in the day of the exam the patients can drink the same clear liquids with or without sugar until 4 hours before the colonoscopy, which will be carried out in the morning).
  Colonoscopy.
  Arms: Dietary supplement
Other: Bowel preparation as usual. — Bowel preparation as usual (one day before the colonoscopy with no ingestion of solid foods, possibly with ingestion of clear liquids with or without sugar (such as tea or other transparent beverages without pulp, but not milk, yogurt, broth or gelatine), and with ingestion of 275,84 g (4 sachets) of polyethylene glycol 3350 (Klean-Prep®) in 4 litres of water in 3 to 4 hours (250 mL every 15 minutes), starting at 18:00; in the day of the exam the patients can drink the same clear liquids with or without sugar until 4 hours before the colonoscopy, which will be carried out in the morning).
  Colonoscopy.
  Arms: Control

SUMMARY:
The high energy nutritional supplement Resource® Energy is approved for human nutritional support in various clinical conditions, yet it has been used off-label to alleviate the effects of hunger during bowel preparation for colonoscopy. Its impact in mucosa visualization quality and hunger alleviation is unknown. The product is liquid and nutritious but it is not transparent, thus it is conceivable that it could alleviate the discomfort of hunger during the preparation but possibly compromising mucosa visualization. In this study, participants who will undergo a colonoscopy (requested for an explicit medical indication) will take two bottles of the nutritional supplement during the usual bowel preparation. The quality of mucosal visualization and the participants opinion regarding satiety and product tolerance during bowel preparation will then be analysed.

DETAILED DESCRIPTION:
The high energy nutritional supplement Resource® Energy is approved for human nutritional support in various clinical conditions. However, it has been recommended by pharmacists to reduce hunger during bowel preparation for colonoscopy, without any medical prescription or recommendation as there is no scientific evidence regarding this use. Its impact in the quality of mucosal visualization during colonoscopy and in relieving hunger is unknown, thus requiring research.

The dietary supplement is liquid and nutritious, each serving consisting of 200 mL containing carbohydrates 42 g, lipids 10 g, proteins 11.2 g and fiber < 1 g, totalling 303 kcal. It is thus conceivable that it can mitigate the discomfortable feeling of hunger during bowel preparation, but because it is not transparent it could possibly hamper mucosa visualization.

One hundred and fifty control patients (with clinical indication for undergoing colonoscopy) will undergo bowel preparation as usual with the standard of care polyethylene glycol 3350 in 4 litres of water (Klean-Prep®): one day before the colonoscopy with no ingestion of solid foods, possibly with ingestion of clear liquids with or without sugar (such as tea or other transparent beverages without pulp, but not milk, yogurt, broth or gelatine), and with ingestion of 275,84 g (4 sachets) of polyethylene glycol 3350 in 4 litres of water in 3 to 4 hours (250 mL every 15 minutes), starting at 18:00; in the day of the exam the patients can drink the same clear liquids with or without sugar until 4 hours before the colonoscopy, which will be carried out in the morning.

One hundred and fifty patients (with clinical indication for undergoing colonoscopy) will undergo bowel preparation as usual and take two servings of Resource® Energy Apricot.

All patients will be asked about feelings of hunger or side effects of bowel preparation and colonoscopy (nausea, vomits, abdominal pain, abdominal discomfort, abdominal pressure, abdominal bloating, syncope, blood in stool, sleep disturbance, work absenteeism) in a scale from 0 to 10, before and after the colonoscopy. This scale is often used to assess appetite.

Colonoscopic mucosa visualization quality will be assessed in all patients using the Boston Bowel Preparation Scale, which is the most thoroughly validated and recommended scale.

Statistical comparison will the be performed between both groups, regarding colonoscopic mucosa visualization and side effects and sensations experienced, such as hunger.

ELIGIBILITY:
Inclusion Criteria:

* individual requesting a non-contraindicated colonoscopy (with clinical indication) at the outpatient clinic.

Exclusion Criteria:

* pregnancy
* Allergy to any ingredient of Resource® Energy Apricot

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2022-05-28 (Actual); Study Completion 2022-05-28 (Actual)

PRIMARY OUTCOMES:
Mucosa visualization quality (Boston Bowel Preparation Scale) | During the procedure
  Mucosa visualization quality assessed using the Boston Bowel Preparation Scale (0 to 9, 0 being the worst)

SECONDARY OUTCOMES:
Adenoma detection rate | During the procedure
  Adenoma detection rate
Amount of rinsing needed | During the procedure
  Amount of water (mL) injected to wash certain areas of the colon
Hunger during bowel preparation | Reported in the day of the procedure
  Self-reported in a scale from 0 to 10 (10 being the worst)

CONTACTS AND LOCATIONS:
Overall Officials: José AS Medeiros, PhD, Study Chair — Clínica de Gastroenterologia
Locations (1):
- Clínica de Gastroenterologia, Coimbra, Coimbra District, Portugal